CLINICAL TRIAL: NCT00856778
Title: Virtue® Male Incontinence Sling Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP001SU
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Stress Urinary Incontinence
Keywords: Male sling; stress urinary incontinence; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Virtue® Male Sling (Other): Subjects implanted with Virtue® Male Sling
  Interventions: Device: Virtue® Male Incontinence Sling

INTERVENTIONS:
Device: Virtue® Male Incontinence Sling — The VIRTUE® male sling is a Class II, implantable, sub-urethral, permanent, non-absorbable support sling indicated for the surgical treatment of male SUI resulting from intrinsic sphincter deficiency. The sling is manufactured from polypropylene and is sold for single use only.

SUMMARY:
This study is a multi-center, global study that will assess the effectiveness and patient satisfaction of the male incontinence sling 12 months after implant as well as the safety profile of the product.

ELIGIBILITY:
Inclusion Criteria:

* Male subject at least 18 yrs old with an estimated life expectancy of more than 5 years
* Confirmed SUI (stress urinary incontinence) through medical history, urodynamics, and/or physical exam
* Subject has completed urodynamics, uroflow, post-void residual and cystoscopy per protocol within 12 months prior to implant
* Subject has intrinsic sphincter deficiency due to one of the following: post-TURP (trans-urethral resection of the prostate), simple open prostatectomy, radical prostatectomy completed at least 6 months prior to implantation date
* Subject is willing to have the Virtue male sling implanted and is able and willing to completed all f/u visits and procedures as indicated in protocol
* Subject agrees to the provisions of the study and has provided written informed consent as approved by the local ethics committee of the respective site

Exclusion Criteria:

* Subject is unable or unwilling to sign the Informed Consent Form and/or comply with provisions of the study
* Subject has active urogenital infection or active skin infection in region of surgery
* Subject has serious bleeding disorders
* Subject has incontinence due to neurogenic causes defined as multiple sclerosis, spinal cord/brain injury,CVA (cerebrovascular accident), detrusor-external sphincter dyssynergia, Parkinson's disease, or similar conditions
* Subject has previous implant to treat SUI
* Subject has undergone radiation, cryosurgery, or brachytherapy to treat prostate or other pelvic cancer with 6 months or is likely to undergo radiation therapy within the next 6 months
* Subject has active urethral or bladder neck stricture disease requiring continued treatment
* Subject has urge predominant incontinence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Comiter, MD, Principal Investigator — Stanford University
Locations (11):
- United States (8):
  - Kaiser Permanente, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Winter Park Urology Associates, Orlando, Florida
  - Northeast Indiana Research, Fort Wayne, Indiana
  - Wayne State University, Dearborn, Michigan
  - NYU Urology Associates, New York, New York
  - McKay Urology, Charlotte, North Carolina
  - University of Texas-M.D. Anderson Cancer Center, Houston, Texas
- Canada (3):
  - Sunybrook Health Sciences Centre, Toronto, Ontario
  - Mortimer S Davis Jewish General Hospital, Montreal, Quebec
  - CHUS Hopital Fleurimont, Sherbrooke, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Implanted With Virtue® Male Sling: The Coloplast Virtue® Male Sling System is a permanent, synthetic suburethral sling, designed for the surgical treatment of male stress urinary incontinence (SUI). The Virtue® sling is made from knitted, monofilament polypropylene, and is for single-use only.
Period: Overall Study
Arm/Group | Subjects Implanted With Virtue® Male Sling
Started | 98
Completed | 74
Not Completed | 24
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 10
Not completed — Study deviation | 2
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Groups:
- Subjects Implanted With Virtue® Male Sling: The Virtue® Male Sling is a Class II, implantable, sub-urethral, permanent, non-absorbable support sling indicated for the surgical treatment of male SUI resulting from intrinsic sphincter deficiency. The sling is manufactured from polypropylene and is sold for single use only.
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 98
Region of Enrollment [Number; unit: participants]
  United States | 62
  Canada | 36

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction Using the Patient Global Impression of Improvement (PGI-I)
Description: Patient satisfaction using the Patient Global Impression of Improvement (PGI-I. Definition of Success: >50% responding "very much better" or "much better".
Time Frame: 12 months post implant
Population: The study was not fully enrolled and therefore underpowered for the planned analyses.
Measure: Number (95% Confidence Interval); unit: % of subjects successful
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 74
% of subjects successful | 41.9 [30.5 to 53.9]

2. Primary Outcome: Assess Change in 24-hour Pad Weight. Definition of Success: >50% With Outcome of Improved, Much Improved, Very Much Improved, or Cured (Dry).
Description: Endpoint definition: Improved = 25-49% reduction of pad weight, Much Improved = 50-89% reduction of pad weight, Very Much Improved = <12 grams or 90% reduction in pad weight, Cured = Dry. Definition of Success: >50% responding "very much better" or "much better".
Time Frame: 12 months
Population: The study was not fully enrolled and therefore underpowered for the planned analyses.
  There are 71 subjects with outcome 2 (pad weight endpoint). Of the 74 with 12 months follow-up, 3 are missing the pad weight improvement assessment.
Measure: Number (95% Confidence Interval); unit: % of subjects successful
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 71
% of subjects successful | 62.0 [49.7 to 73.2]

3. Secondary Outcome: Assess Change in Subject Satisfaction Through ICIQ
Description: The ICIQ-UI Short Form (International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form) is a brief self-assessment instrument applicable to all incontinent patients worldwide that measures the severity of urinary incontinence. The score ranges from 0 to 21 with higher number indicative of worse Urinary Incontinence severity.
Time Frame: Baseline
Population: There are 95 subjects with outcome 3 (ICIQ at baseline). Of the 98 subjects implanted, 3 are missing the baseline ICIQ assessment.
Measure: Mean (Standard Deviation); unit: units on a scale - ICIQ Score
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 95
units on a scale - ICIQ Score | 16.6 (3.2)

4. Secondary Outcome: Assess Change in Subject Satisfaction Through ICIQ
Description: as for outcome 3
Time Frame: 12 months post implant
Population: There are 73 subjects with outcome 4 (ICIQ at 12 months). Of the 74 subjects with 12 months follow-up, 1 is missing the 12 month ICIQ assessment.
Measure: Mean (Standard Deviation); unit: units on a scale - ICIQ Score
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 73
units on a scale - ICIQ Score | 12.0 (6.1)

5. Secondary Outcome: Assess Change in Subject Satisfaction Through the UCLA-RAND Incontinence Index - Urinary Bother
Description: The UCLA-RAND Incontinence Index is from a section within the RAND 36-item Health Survey v2 (SF-36 v2) and UCLA Prostate Cancer Index and measures a patient's urinary habits over the 4 weeks prior to questionnaire completion and consists of 6 questions. Two scores are produced, the Urinary Bother and Urinary Function scores. The Urinary Bother score ranges from 0 to 100 with lower scores indicating worse symptoms of urinary bother. The Urinary Function score ranges from 0 to 100 with lower scores indicating worse urinary function.
Time Frame: Baseline
Population: There are 97 subjects with outcome 5 (Urinary bother at baseline). Of the 98 subjects implanted, 3 are missing the baseline Urinary Bother assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 97
units on a scale | 13.7 (20.7)

6. Secondary Outcome: Assess Change in Subject Satisfaction Through the UCLA-RAND Incontinence Index - Urinary Bother
Description: as for outcome 5
Time Frame: 12 months post implant
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 74
units on a scale | 36.5 (34.9)

7. Secondary Outcome: Assess Change in Subject Satisfaction Through the UCLA-RAND Incontinence Index - Urinary Function
Description: as for outcome 5
Time Frame: Baseline
Population: There are 97 subjects with outcome 7 (Urinary function at baseline). Of the 98 subjects implanted, 1 is missing the baseline Urinary Function assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 97
units on a scale | 17.1 (12.6)

8. Secondary Outcome: Assess Change in Subject Satisfaction Through the UCLA-RAND Incontinence Index - Urinary Function
Description: as for outcome 5
Time Frame: 12 months post implant
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 74
units on a scale | 37.1 (28.2)

9. Secondary Outcome: Assess Change in Pad Use
Description: Patients reported the average number of pads used in a 24 hour period over the 4 weeks prior to the assessment.
Time Frame: Baseline
Population: There are 97 subjects with outcome 9 (baseline pad use). Of the 98 subjects implanted, one is missing the baseline assessment of pad use.
Measure: Mean (Standard Deviation); unit: pads/24 hours
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 97
pads/24 hours | 4.1 (3.6)

10. Secondary Outcome: Assess Change in Pad Use
Time Frame: 12 months post-implant
Measure: Mean (Standard Deviation); unit: pads/24 hours
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 74
pads/24 hours | 2.4 (2.1)

11. Secondary Outcome: Physician Questionnaire - Virtue® Surgical Procedure Was Straightforward
Time Frame: At implant
Measure: Number; unit: percentage of responses
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 98
percentage of responses
  Strongly disagree | 4.1
  Somewhat disagree | 6.1
  Neutral | 3.1
  Somewhat agree | 24.5
  Strongly agree | 62.2

12. Secondary Outcome: Physician Questionnaire - Virtue® Procedure Was as Easy as Competitive Therapies
Time Frame: At implant
Measure: Number; unit: percentage of responses
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 98
percentage of responses
  Strongly disagree | 3.1
  Somewhat disagree | 13.3
  Neutral | 10.2
  Somewhat agree | 9.2
  Strongly agree | 64.3

13. Secondary Outcome: Physician Questionnaire - Virtue® Was Easy to Position Over the Bulbous Urethra
Time Frame: At implant
Measure: Number; unit: percentage of responses
Arm/Group | Subjects Implanted With Virtue® Male Sling
Number analyzed (Participants) | 98
percentage of responses
  Strongly disagree | 3.1
  Somewhat disagree | 2.0
  Neutral | 3.1
  Somewhat agree | 30.6
  Strongly agree | 61.2

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Subjects Implanted With Virtue® Male Sling
Serious Adverse Events (participants affected / at risk) | 2/98
Other Adverse Events (participants affected / at risk) | 26/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Implanted With Virtue® Male Sling (N=98)
Hematoma (Surgical and medical procedures) | 1 (1)
Urosepsis (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Implanted With Virtue® Male Sling (N=98)
Paresthesia (genital) (Surgical and medical procedures) | 12 (12)
Perineal pain (Surgical and medical procedures) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No